CLINICAL TRIAL: NCT04549389
Title: Comparing 2 Frequency Protocols of Low-intensity Shockwave Therapy for Non-bacterial Chronic Prostatitis Type IIIb /Chronic Pelvic Pain Syndrome: a Randomised Clinical Trial
Brief Title: The Ideal LiST Session Frequency Protocol for CPPS Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases Theesaloniki, Greece, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1410/2020
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pelvic Pain Syndrome; Chronic Non-bacterial Prostatitis Type IIIB

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive 6 Low-intensity shockwave therapy (LiST) sessions (1/week) by using Dornier Aries 2 shockwave machine (energy level 7)
  Interventions: Device: Low intensity shockwave therapy
- Group B (Active Comparator): Patients will receive 6 Low-intensity shockwave therapy (LiST) sessions (2/week) by using Dornier Aries 2 shockwave machine (energy level 7)
  Interventions: Device: Low intensity shockwave therapy

INTERVENTIONS:
Device: Low intensity shockwave therapy — LiST will be applied in the perineum of the patients by using Dornier Aries 2 shockwave machine (5000shockwaves per session, energy level 7)

SUMMARY:
The study will include 50 chronic pelvic pain syndrome (CPPS) patients who will be randomised in 2 groups.

Group A (25 patients )will receive 6 LiST sessions with a frequency 1 session / week.

Group B (25 patients) will receive 6 LiST sessions with a frequency 2 sessions / week.

National Institutes of Health Chronic Prostatitis Symptom Index(NHI-CPSI), International Prostate Symptom Score (IPSS), International Index of Erectile Function (IIEF-ED) questionnaires will be answered before and at 1 and 3 month follow up visit.

Adverse events will be reported during the treatment and follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must 18 to 60 years of age.
2. Participant has signed and dated the appropriate Informed Consent document.
3. Participant has had a clinical diagnosis of CP/CPPS defined as symptoms of discomfort or pain in the perineal or pelvic region for at least a three (3) month period within the last six (6) months

Exclusion Criteria:

1. Participant has evidence of facultative Gram negative or enterococcus with a value of ≥ 1000 CFU/ml in mid-stream urine (VB2).
2. Participant has a history of prostate, bladder or urethral cancer.
3. Participant has undergone pelvic radiation or systemic chemotherapy.
4. Participant has undergone intravesical chemotherapy.
5. Participant has unilateral orchialgia without pelvic symptoms, active urethral stricture or bladder stones, or any other urological condition associated with LUTS, any neurological disease or disorder affecting the bladder.
6. Participant has undergone prostate surgery or treatment.
7. Participant with penile or urinary sphincter implants.
8. Participant has been diagnosed with cancer during the last 5 years, or had any surgery in the pelvis.
9. Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.
10. PSA>3 and age > 40 years
11. Positive (suspicious for malignancy) digital rectal examination (DRE).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
1.The difference between groups in the change of the pain domain of NIH-CPSI score | from baseline to 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special pain domain (items 1-4) and the score for this domain ranges from 0 to 21.

SECONDARY OUTCOMES:
The difference between groups in the change of total NIH-CPSI score (Q1-9) | Time Frame: baseline, 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome)
The difference between groups in the change of urinary symptoms (Q 5-6) and quality of life domains (Q 7-9) of the NIH-CPSI score | from baseline to 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special urinary symptom domain (items 5-6) and the score for this domain ranges from 0 to 10
The difference between groups in the change of IIEF-ED score | from baseline to 4 and 12 weeks after final treatment
  It will be assessed by International Index of Erectile Function -Erectile Domain (IEF-ED) score. A questionnaire designed to evaluate erectile capabilities. The questionnaire provides a score between 5 and 30.The severity categories are: 1-10 severe ED, 10-16 moderate ED, 17-21 moderate to mild ED, 22-25 mild ED, 26-30 no ED
The difference between groups in the change of IPSS | from baseline to 4 and 12 weeks after final treatment
  They will be assessed by the International Prostate Symptom Score (IPSS). A questionnaire designed to provide information on lower urinary tract symptoms and their impact on quality of life. Scores range from 0 to 35. The severity categories are: 1-7 mild, 8-19 moderate, 20-35 severe
The difference between groups in the the Pain Visual Analogue Scale (VAS) | at week 3, 4, 5,
  It will be assessed by the pain VAS, right after each LIST session. Pain VAS is a unidimensional measure of pain intensity . It is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]. To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm)
Adverse events rate in all patients | 18 weeks
  Potential treatment related adverse events after the first LIST session and during the 3 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Professor, Principal Investigator — Institute for the Study of Urological Diseases, Thessaloniki, Greece
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No